CLINICAL TRIAL: NCT06233877
Title: An Open Label Phase 2 Trial to Evaluate the Safety, Tolerability, and Efficacy of Low Dose G-FLIP in Combination With Mitomycin C in Patients With Stage IV Pancreatic Cancer Who Have Failed First-Line Treatment
Brief Title: Clinical Trial Evaluating Low Dose G-FLIP Plus Mitomycin C for Stage IV Pancreatic Cancer
Acronym: GFLIPM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hirschfeld Oncology (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-FLIP-M Pancreatic
Record Dates: First submitted 2024-01-10; First posted 2024-01-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic; low dose
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- G-GLIP plus Mitomycin C (Experimental): G-FLIP: Gemcitabine, Fluorouracil, Leucovorin, Irinotecan, and Oxaliplatin every 2 weeks plus Mitomycin C every 4 weeks
  Interventions: Drug: G-GLIP plus Mitomycin C

INTERVENTIONS:
Drug: G-GLIP plus Mitomycin C — G-FLIP: Gemcitabine, Fluorouracil, Leucovorin, Irinotecan, and Oxaliplatin plus Mitomycin C

SUMMARY:
The study focuses on advanced metastatic pancreatic cancer, testing a combination of low-dose anti-cancer drugs (G-FLIP: Gemcitabine, Fluorouracil, Leucovorin, Irinotecan, and Oxaliplatin) with the addition of Mitomycin C. The aim is to find a safer and more effective therapy for this devastating disease.

DETAILED DESCRIPTION:
Objective: Evaluate the safety, tolerability, and efficacy of G-FLIP combined with Mitomycin C for advanced pancreatic cancer.

Design: Open-label study with 60 evaluable subjects. Treatments: G-FLIP administered every 2 weeks, with Mitomycin administered every 4 weeks.

Efficacy Assessments: Based on response criteria (Complete Response, Partial Response, Stable Disease, Progressive Disease), Response Rate, Progression-Free-Survival, Overall Survival, and 12-Month Survival Rate.

Safety Assessments: Include physical exams, symptom evaluation, vital signs, ECOG performance status, clinical pathology, urinalysis, and Quality of Life assessments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic (Stage IV) pancreatic adenocarcinoma.

  * Failed first-line chemotherapy.
  * ECOG performance status of 0-2.
  * Expected survival of more than 3 months.
  * Adequate organ function as indicated by lab values.
  * Age 18 or older.
  * Signed informed consent.

Exclusion Criteria:

* • Known brain metastases.

  * Significant cardiovascular or other uncontrolled diseases.
  * Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Baseline, 3 months, 6 months, 1 year, and then annually up to 5 years.
  This measure assesses the duration of time from the start of the study until death from any cause.
Response Rate | Baseline, 3 months, 6 months, 1 year, and then annually up to 5 years.
  This measure assesses the rate of disease progression or worsening, as determined by changes in tumor size and appearance on radiological scans. The evaluation is conducted using the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, which provide a standardized method for measuring tumor size and categorizing response to treatment."

CONTACTS AND LOCATIONS:
Locations (1):
- Hirscheld Oncology, Brooklyn, New York, United States